CLINICAL TRIAL: NCT06752642
Title: Conventional Denture Versus Implant Overdenture Opposing Mandibular Implant Overdenture: Residual Alveolar Bone Height Changes of the Premaxilla
Brief Title: CD vs IOD Opposing Mandibular IOD : Bone Height Changes of the Premaxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Moataz Mohamed Soliman Elezaby, PhD researcher, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M01030821
Record Dates: First submitted 2024-11-28; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Edentulism
Keywords: overdenture; implants; maxilla; edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxillary conventional denture and mandibular implant overdenture (Active Comparator): Participants have maxillary complete denture opposing mandibular implant overdenture
  Interventions: Procedure: Implant overdenture
- maxillary and mandibular implant overdenture (Active Comparator): Participants have maxillary implant overdenture opposing mandibular implant overdenture
  Interventions: Procedure: Implant overdenture

INTERVENTIONS:
Procedure: Implant overdenture — patients received implant overdenture

SUMMARY:
The goal of this clinical trial is to evaluate bone resorption of the anterior region of maxillary arch. The main questions it aims to answer are:

Does implants assisting maxillary complete denture enhance stability, retention and mastication of the patient ?

Does implants assisting maxillary complete denture reduce bone resorption in the anterior region of maxilla ?

Participants will:

* receive 2 implants with attachments assisting their maxillary complete denture
* Visit the clinic once every 6 months for checkups and tests

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation.

The trial will include A total of twenty male adult patients unsatisfied with their maxillary complete denture seeking to enhance their mastication and esthetics. The participants will be recruited from the Outpatient clinic at Faculty of Dentistry, Mansoura University.

each patient will receive 2 implants with attachments to assist their maxillary complete denture then follow up every 6 months for checkups.

No active advertisement will be used for participant recruitment, and instead, a convenience sample will be formed. Prior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The protocol of the study was approved by Mansoura University's ethics committee before initiation

ELIGIBILITY:
Inclusion Criteria:

1. General good health without any systemic diseases affecting bone resorption such as uncontrolled diabetes or osteoporosis. This was confirmed through taking medical history and clinical examination by a physician.
2. Having angel's class I maxillo-mandibular relationships.
3. Presence of sufficient bone quality and quantity in the anterior region of maxilla and mandible which allow inserting implants of at least 3.75 mm diameter and 10 mm length. This was verified by Preoperative low dose Cone Beam (C.T) d) Presence of sufficient restorative space (a minimum of 15 mm must be available from the mucosa covering the crest of the residual ridge to the proposed occlusal plane), this was confirmed by tentative jaw relation.

(e) Having maladaptive maxillary conventional complete denture.

Exclusion Criteria:

1. Uncontrolled systemic diseases such as: uncontrolled hypertension, or uncontrolled cardiovascular disease
2. metabolic disorders such as diabetes mellitus
3. Patients with compromised immune systems as (Long term immunosuppressant and corticosteroid drug
4. TMJ dis orders and neuromuscular diseases
5. Patient with abnormal habits as clenching and bruxism, Smoking patient, Uncooperative patients.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
bone height changes | 18 months
  assessment of bone height changes in the premaxilla

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M. Elezaby, PhD student, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No